CLINICAL TRIAL: NCT03438331
Title: Effects of Group Cognitive Behavioural Therapy on Comorbid Insomnia and Depression in Youth: a Randomised, Assessor Blind, Parallel Group Trial
Brief Title: Effects of Group Cognitive Behavioural Therapy on Comorbid Insomnia and Depression in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Chinese University of Hong Kong (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Dr. Shirley Xin Li, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27613017
Record Dates: First submitted 2018-01-02; First posted 2018-02-19 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Insomnia; Depression
Keywords: Insomnia; Depression; Adolescents; Youth
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CBT-I (Experimental)
  Interventions: Behavioral: Cognitive Behavioural Therapy for Insomnia (CBT-I)
- CBT-D (Active Comparator)
  Interventions: Behavioral: Cognitive Behavioural Therapy for Depression (CBT-D)
- Waiting-list control (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive Behavioural Therapy for Insomnia (CBT-I) — The intervention will consist of 8 weekly group sessions (90-min, 5-8 adolescents in each group) of CBT-I delivered within a 10-week window. The treatment components in the CBT-I aim to address the behavioural, cognitive and physiological perpetuating factor of insomnia and include: psycho-education about sleep and sleep hygiene, stimulus control, sleep restriction, relaxation training, structured worry time, cognitive restructuring (targeting sleep-related dysfunctional cognitions), and relapse prevention.
  Arms: CBT-I
Behavioral: Cognitive Behavioural Therapy for Depression (CBT-D) — The intervention will consist of 8 weekly group sessions (90-min, 5-8 adolescents in each group) of CBT-D delivered within a 10-week window. The main treatment elements of CBT-D include: psycho-education about depression, self-monitoring, behavioural activation, improving social skills, communication skills and problem solving skills, cognitive restructuring (addressing negative and irrational thoughts often associated with depression in adolescents), relaxation techniques, and relapse prevention.
  Arms: CBT-D

SUMMARY:
Major depressive disorder (MDD) is among the most common psychiatric disorders among adolescents, and is associated with considerable psychosocial and functional impairments and an elevated risk of suicidal behaviour and completed suicide. Meanwhile, sleep disturbance, particularly insomnia, is among the most prevalent and prominent presenting complaints in adolescents with depression. Despite its high prevalence, insomnia often remains overlooked and under-treated in clinical practice. However, growing evidence suggests an intricate relationship between insomnia and depression, which has become an area in need of further focused attention. This project will involve a randomised controlled trial proposed to examine whether insomnia treatment confers additional benefit to depression treatment in adolescents with comorbid depression and insomnia, for improving sleep and depressive symptoms, and other clinical and daytime symptoms as well as overall functional improvement in both the short and long term. Eligible adolescent participants will be randomised to either intervention (8-week group Cognitive Behavioural Therapy for Insomnia, CBT-I, or 8-week group Cognitive Behavioural Therapy for Depression, CBT-D) or waiting-list control condition. Assessments will be conducted at pre-treatment (week 0), during the treatment (week 2, 4, 6) and post-treatment (week 8/at the conclusion of the last group session). The two active treatment groups will be additionally followed up at posttreatment one-month and six-month.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese aged 12-24 years old;
2. Written informed consent of participation into the study is given by the participant and his/her parent or guardian (for those aged under 18);
3. Being able to comply with the study protocol;
4. Having a DSM-V diagnosis of insomnia disorder, with a score on Insomnia Severity Index (ISI) >=9; AND a DSM-V diagnosis of depressive disorder

Exclusion Criteria:

1. A current diagnosis of substance abuse or dependence; a current or past history of manic or hypomanic episode, schizophrenia spectrum disorders, neurodevelopmental disorders, organic mental disorders, or intellectual disabilities;
2. Having a prominent medical condition known to interfere with sleep continuity and quality (e.g. eczema, gastro-oesophageal reflux disease);
3. Having a clinically diagnosed sleep disorder that may potentially contribute to a disruption in sleep continuity and quality, such as narcolepsy, sleep-disordered breathing, and restless leg syndrome, as ascertained by DISP;
4. Concurrent, regular use of medications(s) known to affect sleep continuity and quality (e.g. hypnotics, steroids);
5. In the opinion of the research clinician, having a clinically significant suicidality (presence of suicidal ideation with a plan or an attempt);
6. Having been enrolled in any other clinical trial investigational products within one month at the entry of the study;
7. Initiation of or change in antidepressant medication within past 2 months;
8. Having been or is currently receiving any structured psychotherapy;
9. With hearing or speech deficit;
10. Night shift worker.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 133 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
Change of depressive symptoms (assessor-rated) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Children's Depression Rating Scale (CDRS-R) is a 17-item rating scale based on a semistructured interview with children. Possible scores range from 17 to 113, with higher scores indicating severer depressive symptoms.
Change of self-report mood symptoms | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Hospital Anxiety and Depression Scale (HADS) is a self-assessed scale for detecting states of depression and anxiety. The depression subscale range in scores from 0 to 21, with higher scores indicating severer states of depression. Similarly, the anxiety subscale range in scores from 0-21 with higher scores indicating severer states of anxiety. No additional computation will be made with the two subscores.
Change of insomnia symptoms | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Insomnia Severity Index (ISI) is a 5-item self-rated scale. Possible scores range from 0 to 20, with higher scores indicating higher insomnia severity.

SECONDARY OUTCOMES:
Change of sleep quality | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Pittsburgh Sleep Quality Index (PSQI) is a self-rated scale consisting of 19 questions. All items are combined to form seven component scores on different aspects of sleep quality, each of which ranges from 0 to 3 points with higher scores representing more sleep disturbance. The seven component scores are added to one global score, which ranges from 0 to 21, with higher scores indicating more difficulties with sleep.
Change of sleep diary measure (time in bed, TIB) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: time in bed (TIB) in hours
Change of sleep diary measure (total sleep time, TST) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: total sleep time (TST) in hours
Change of sleep diary measure (sleep onset latency, SOL) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep onset latency (SOL) in mins
Change of sleep diary measure (wake after sleep onset, WASO) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: wake after sleep onset (WASO) in mins
Change of sleep diary measure (sleep efficiency, SE) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Daily sleep diary for consecutive seven days. Sleep parameter estimated by daily sleep diary: sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %
Change of objective sleep measure (time in bed, TIB) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: time in bed (TIB) in hours
Change of objective sleep measure (total sleep time, TST) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: total sleep time (TST) in hours
Change of objective sleep measure (sleep onset latency, SOL) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: sleep onset latency (SOL) in mins
Change of objective sleep measure (wake after sleep onset, WASO) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: wake after sleep onset (WASO) in mins
Change of objective sleep measure (sleep efficiency, SE) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Actigraphic assessment for consecutive seven days. Sleep parameter estimated by wrist actigraphy: sleep efficiency (SE), which is calculated by total sleep time divided by total time in bed, %
Change of daytime sleepiness | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Paediatric Daytime Sleepiness Scale (PDSS) is an 8-item self-rated scale measuring daytime sleepiness, ranging in total scores from 0 to 32 with higher scores indicating more sleepiness.
Change of daytime fatigue | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Multidimensional Fatigue Inventory (MFI) is a 20-item self-rated scale on fatigue symptoms. There are three subscales, measuring the physical (possibly scored from 7 to 35), mental (possibly scored from 6 to 30), and spiritual (possibly scored from 7 to 35), dimensions of fatigue. A grand total score can be calculated by summing up the three sub scores. In all cases, a higher score represents higher fatigue symptoms.
Change of quality of life | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  KIDSCREEN-27 is a 27-item self-rated scale measuring health related quality of life measure for children and adolescents. There are five subscales on: physical well-being (possibly scored from 5 to 25), psychological well-being (possibly scored 7 to 35), autonomy & parents (possibly scored 7 to 35), peers & social support (possibly scored 4 to 20), and school environment (possibly scored 4 to 20). A grand total score can be calculated by summing up the five sub scores. In all cases, a higher score represents higher perceived well-being.
Change of suicidal ideation | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Depressive Symptom Inventory Suicidality Subscale (DSI-SS) is a 4-item self-rated scale measuring suicidal ideation. Possible total scores range from 0 to 12, with higher scores indicating higher suicidal ideation.
Change of subjective cognitive performance | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Cognitive Failures Questionnaire (CFQ) is a 20-item self-rated scale measuring perceived failures in daily cognitive tasks. Possible total scores range from 0 to 80, with higher scores indicating higher cognitive failures.
Change of objective cognitive performance (visual attention & task switching) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Trail Making Test for assessing visual attention and task switching. In Trail Making Test, longer reaction time indicates lower level of attention.
Change of objective cognitive performance (inhibitory ability) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Go/No-go Task for assessing inhibitory ability. In Go/No-go Task, a higher error rate indicates lower inhibition control.
Change of objective cognitive performance (working memory by digit span) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Digit Span Task for assessing working memory capacity. In Digit Span Task, a higher number of recalled digits indicates better working memory.
Change of objective cognitive performance (working memory by N-Back) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  N-back Task for assessing working memory capacity and manipulation. In N-back Task, a d prime score will be calculated based on the signal detection theory, where a higher score indicates better working memory performance.
Change of objective cognitive performance (episodic memory) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Chinese Auditory Verbal Learning Task for assessing episodic memory, where a higher number of recalled words indicates better episodic memory performance.
Change of objective cognitive performance (problem solving) | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Wisconsin Card Sorting Test for assessing problem solving. In Wisconsin Card Sorting Test, lower executive functioning is indicated by a higher percentage of persistent errors and a higher number of trials taken to complete the first category.
Change of sleep related attention bias | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Sleep-related Dot-Probe Task for assessing sleep-related attention bias. In the Sleep-related Dot-probe Task, a higher attention bias score indicates higher vigilance towards sleep-related stimuli.
Change of risk-taking & decision making | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month and six-month for those in the two active treatment groups
  Balloon Analogue Risk Task for assessing risk-taking and decision-making. In Balloon Analogue Risk Task, a score will be calculated by averaging the number of pumps on unexploded blue balloons, where a higher score indicates more risk-taking and impulsive propensities.
Change of dysfunctional beliefs and attitudes about sleep | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Dysfunctional Beliefs and Attitudes about Sleep (DBAS) is a 16-item self-rated scale measuring the respondent's sleep-related beliefs, more specifically, their expectations and attitudes regarding the causes, consequences, and potential treatments of sleep issues. A total score is calculated by averaging score of all items, possibly scored 0 to 10, with a higher score indicating more dysfunctional beliefs and attitudes about sleep.
Change of sleep hygiene and practice | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Sleep Hygiene Practice Scale (SHPS) is a 30-item self-rated scale measuring sleep hygiene behaviors, ranging in total scores from 30 to 180, with higher scores indicating lower levels of sleep hygiene.
Change of pre-sleep arousal | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Pre-Sleep Arousal Scale is a 16-item self-rated scale measuring pre-sleep arousal. There are two subscales on the cognitive and somatic manifestations of arousal, with eight items in each subscale (possibly scored from 8 to 40). In both cases, a higher score indicates higher pre-sleep arousal.
Change of overall severity of clinical symptoms | Baseline, post-treatment (week 8/at the conclusion of last group session) for all participants; and additionally at post-treatment one-month, six-month and 24-month for those in the two active treatment groups
  Clinical Global Impression (CGI) Scale is a clinician-rated scale, comprised of two one-item subscales: Severity of Illness (CGI-S) subscale evaluating the severity of psychopathology, and Clinical Global Improvement Scale (CGI-I) evaluating change from the initiation of treatment. In both cases, the score is given on a seven-point scale, with higher values indicating higher severity of illness and larger improvement respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Xin Li, PhD,DClinPsy, Principal Investigator — The University of Hong Kong
Locations (1):
- Sleep Research Clinic & Laboratory, Department of Psychology, The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No